CLINICAL TRIAL: NCT00659386
Title: Intravenous Immunoglobulin Therapy for Patients With Idiopathic Cardiomyopathy and Endomyocardial Biopsy Proven High PVB19 Viral Load
Brief Title: IVIg Therapy for Patients With Idiopathic Cardiomyopathy and Endomyocardial Biopsy Proven High PVB19 Viral Load
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: S. Heymans, Maastricht UMC+
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: MEC 08-4-010
Record Dates: First submitted 2008-04-07; First posted 2008-04-16 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Heart Failure
Keywords: Heart failure; Parvovirus B19; Intravenous immuneglobulin
MeSH Terms: conditions — Heart Failure | interventions — gamma-Globulins; Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Patients with chronic idiopathic cardiomyopathy and EMB proven high PVB19 virus load.
  Interventions: Drug: Intravenous immunoglobulin therapy

INTERVENTIONS:
Drug: Intravenous immunoglobulin therapy — Patients received total dose of 2 g/kg of immune globulin administered as 0.5 g/kg IV over a period of 6 hours on each of 3 consecutive days.
  Other Names: IVIG

SUMMARY:
Rationale: Parvovirus B19 (PVB19) persistence in the heart has been associated with progressive cardiac dysfunction and evolution to dilated cardiomyopathy.

Objective: Whether high dose of intravenous immunoglobulin (IVIg) in addition to conventional heart failure therapy achieves virus reduction, thereby resulting in improvement of cardiac function.

Study design: A interventional study of virus presence and cardiac functional capacity before and after IVIg therapy.

Study population: Patients with idiopathic cardiomyopathy and symptomatic heart failure for more than 1 year and a significant PVB19 viral load in endomyocardial biopsies (EMB) and treated with high dose of IVIg were included.

Intervention (if applicable): Patients were treated with a total dose of 2 g/kg of immune globulin administered as 0.5 g/kg IV over a period of 6 hours on each of 4 consecutive days.

Main study parameters/endpoints: EMBs: virus (PVB19, enteroviruses, adenoviruses, Epstein-Barr virus, human herpes virus-6 and cytomegalovirus), inflammation (lymphocytes an macrophages) and fibrosis. Cardiac functional capacity: NYHA classification, echocardiographic evaluation (left ventricular ejection fraction, end-systolic diameter, end-diastolic diameter).

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic heart failure <1 year.
* Optimal conventional heart failure medication <6 months.
* PVB19 viral load >150copies/mcg DNA in EMBs.

Exclusion Criteria:

* significant (lesions >50% stenosis) coronary artery disease.
* significant valvular disease.
* systemic diseases such as sarcoidosis, giant cell myocarditis, hemochromatosis, or systemic autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-02 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
viral loads in EMBs before and after therapy | At baseline and 6 month follow-up

SECONDARY OUTCOMES:
Echocardiographic analysis, NYHA functional class, type/degree of inflammation and fibrosis in the myocardium. | at baseline and at 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Heymans, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- University Hospital Maastricht, Maastricht, Maastricht, Netherlands

REFERENCES:
- [Derived] Dennert R, Velthuis S, Schalla S, Eurlings L, van Suylen RJ, van Paassen P, Tervaert JW, Wolffs P, Goossens VJ, Bruggeman C, Waltenberger J, Crijns HJ, Heymans S. Intravenous immunoglobulin therapy for patients with idiopathic cardiomyopathy and endomyocardial biopsy-proven high PVB19 viral load. Antivir Ther. 2010;15(2):193-201. doi: 10.3851/IMP1516. PMID 20386074